CLINICAL TRIAL: NCT05463328
Title: Open Versus Laparoscopic Assisted Pancreaticoduodenectomy: Randomized Control Comparative Prospective Study
Brief Title: Open Versus Laparoscopic Assisted Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Aly, assistant lectuerer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pancreaticoduodenectomy
Record Dates: First submitted 2022-04-08; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Pancreas Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic assisted pancreaticoduodenctomy (Experimental): If inclusion criteria are met ,these group of patients will undergo Laparoscopic assisted pancreaticoduodenctomy.
  Interventions: Procedure: laparoscopic assisted pancreaticoduodenectomy
- Open pancreaticduodenctomy (Active Comparator): criteria are met ,these group of patients will undergo open pancreaticoduodenctomy
  Interventions: Procedure: Open pancreaticduodenctomy

INTERVENTIONS:
Procedure: laparoscopic assisted pancreaticoduodenectomy — laparoscopic assisted pancreaticoduodenectomy.
  Arms: Laparoscopic assisted pancreaticoduodenctomy
Procedure: Open pancreaticduodenctomy — Open pancreaticduodenctomy
  Arms: Open pancreaticduodenctomy

SUMMARY:
Compare open and laparoscopic assisted pancreaticoduodenectomy regarding intraoprative blood loss, organ injury, completion of planned laparoscopic steps, duration and early post operative course of pain, hem stability, oral feeding, leakage(pancreatic, billary and intestinal). ,bleeding, mortality, lymph nodes and safety margins .

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is the only option curative intended in the treatment of resectable pancreatic ductal adenocarcinomas, duodenal carcinoma, ampullary carcinoma, lower common bile duct cholangiocarcinoma,. It is still associated with very high morbidity and mortality. [1]. Pancreatic cancer ranks as the seventh leading cause of cancer-related death worldwide, and the fourth among other cancers[2,3]. In recent years, the minimally invasive techniques has considered revolution in surgeries of pancreatic cancers [4,5]. Laparoscopic assisted pancreaticoduodenectomy is a hybrid procedure combining laparoscopic resection and reconstruction through a small incision.it companies laparoscopic mobilization and dissection due to magnification compared with open pancreaticoduodenectomy[6]. Several studies have shown that laparoscopic assisted pancreaticoduodenectomy could result in less blood loss less, pain ,less wound infection and shorter hospital stay compared to open pancreaticoduodenectomy[7,8]. Limited literature described the safety and efficacy of laparoscopic assisted pancraticododenostomy .Also such comparative studies deficient in evaluation of outcomes of laparoscopic assisted pancraticododenostomy and open pancraticoduodenoctomy.So the interest of our study is to compare between the feasibility and safety of laparoscopic assisted pancraticododenostomy and open pancraticoduodenoctomy.

ELIGIBILITY:
Inclusion Criteria:

1. age less than 70 years.
2. resectable tumour,
3. fit for surgery

Exclusion Criteria:

1. patients with jaundice with serum bilirubin above 200mml/dl.
2. patients with bleeding tendency until corrected.
3. patients with advanced and metastatic malignancy.
4. patients with cardiopulmonary diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
post operative pain. | Compare the post operative pain between open and laparoscopic assisted pancreaticoduodenctomy in the first week after operation
  Compare the post operative pain betweenopen and laparoscopic assisted pancreaticoduodenectomy
Blood loss | Compare the intra operative blood loss between open and laparoscopic assisted pancreaticoduodenectomy during the operation
  Compare between the intra operative blood loss in the open and laparoscopic assisted pancreaticoduodenectomy
Rate of postoperative anastomosis leakage(pancreatic,billary and intestinal). | Rate of postoperative anastomosis leakage(pancreatic,billary and intestinal) in the first month after operation
  Compare the rate of postoperative anastomosis leakage(pancreatic,billary and intestinal) between the open and laparoscopic assisted pancreaticoduodenctomy

SECONDARY OUTCOMES:
Postoperative haemorrhage | In the first 2 weeks
  Compare between the postoperative haemorrhage by cc in the open and laparoscopic assisted pancreaticoduodenectomy
Postoperative wound infection. | In the first 2 weeks
  Compare between the postoperative wound infection in the open and laparoscopic assisted pancreaticoduodenectomy
Starting oral feeding | In the first 3 days after operation
  Compare between starting oral feeding in the open and laparoscopic assisted pancreaticoduodenectomy
Postoperative 30 days mortality rate. | In the first 30days after operation
  Compare between the Postoperative 30 days mortality rate in the open and laparoscopic assisted pancreaticoduodenectomy

REFERENCES:
- [Background] Newhook TE, LaPar DJ, Lindberg JM, Bauer TW, Adams RB, Zaydfudim VM. Morbidity and mortality of pancreaticoduodenectomy for benign and premalignant pancreatic neoplasms. J Gastrointest Surg. 2015 Jun;19(6):1072-7. doi: 10.1007/s11605-015-2799-y. Epub 2015 Mar 24. PMID 25801594
- [Background] Erratum to "Cancer statistics, 2021". CA Cancer J Clin. 2021 Jul;71(4):359. doi: 10.3322/caac.21669. Epub 2021 Apr 19. No abstract available. PMID 34232515
- [Background] Correction to Lancet Gastroenterol Hepatol 2019; 4: 934-47. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):e2. doi: 10.1016/S2468-1253(20)30018-2. No abstract available. PMID 32061329
- [Background] Bausch D, Keck T. Minimally Invasive Surgery of Pancreatic Cancer: Feasibility and Rationale. Visc Med. 2018 Dec;34(6):440-443. doi: 10.1159/000495324. Epub 2018 Nov 28. PMID 30675490